CLINICAL TRIAL: NCT06749184
Title: Determining Factors That Predict Hypotension Related to Spinal Anesthesia in Patients With Hypertension
Brief Title: Predictors of Spinal Anesthesia-Induced Hypotension in Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 3.05.2024-27769
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Spinal Anesthesia-Induced Hypotension
Keywords: Spinal Anesthesia; Hypotension; Hypertensive Patients; Hemodynamic Predictors
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to evaluate predictive factors for spinal anesthesia-induced hypotension (SASH) in hypertensive patients undergoing elective surgery. Parameters such as internal jugular vein collapsibility index, carotid intima-media thickness, and flow-mediated dilation will be assessed using ultrasonography to determine their association with SASH. Demographic, anthropometric, and hemodynamic data will also be analyzed. The findings may improve perioperative management strategies for hypertensive patients receiving spinal anesthesia.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between carotid intima-media thickness (CIMT) and spinal anesthesia-induced hypotension (SASH) in hypertensive patients. SASH is a common side effect of spinal anesthesia, with an incidence ranging from 15% to 33%, and is associated with significant clinical consequences such as increased morbidity and mortality. CIMT is a well-established marker of atherosclerotic burden and cardiovascular risk. This study hypothesizes that CIMT may be an independent predictor of SASH in hypertensive patients. Participants will undergo preoperative CIMT measurements and standardized spinal anesthesia procedures, with hemodynamic variables and potential risk factors recorded for analysis.

ELIGIBILITY:
Inclusion Criteria:

Adult hypertensive patients classified as ASA II-III risk group. Patients scheduled for elective surgeries requiring spinal anesthesia.

Exclusion Criteria:

Presence of severe renal or hepatic failure, or severe respiratory or cardiovascular diseases.

Contraindication to spinal anesthesia. Failure of spinal anesthesia. History of carotid surgery or presence of carotid plaques. Presence of anxiety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult hypertensive patients scheduled for elective surgical procedures under spinal anesthesia at Konya City Hospital. The target population comprises patients with hypertensive patients (ASA II-III classification), who are deemed fit for elective surgery and spinal anesthesia by their clinical teams.
  Eligible participants will be screened based on inclusion and exclusion criteria. The study population represents a subset of hypertensive individuals with varying durations of hypertension, medication regimens, and cardiovascular profiles. Patients will be recruited from preoperative assessment clinics and surgical wards at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Spinal Anesthesia-Induced Hypotension (SASH) | 30 minutes after spinal anesthesia.
  Percentage of patients experiencing a decrease in systolic blood pressure by 20% or more from baseline or a drop below 90 mmHg during the first 30 minutes following spinal anesthesia.

OTHER OUTCOMES:
Predictive Value of Internal Jugular Vein Collapsibility Index | Pre-anesthesia measurement.
  The collapsibility index of the inferior vena cava (IVC) will be measured using ultrasound. Measurements will be obtained during inspiration and expiration, and the collapsibility index will be calculated as [(IVC diameter during expiration - IVC diameter during inspiration) / IVC diameter during expiration] × 100%. Measurements will be performed preoperatively and 30 minutes after spinal anesthesia induction.
Flow-Mediated Dilation (FMD) | Pre-anesthesia measurement.
  FMD will be measured using high-resolution ultrasound to assess endothelial function. Measurements will be performed on the brachial artery at baseline and after inducing hyperemia with a blood pressure cuff. FMD will be calculated as [(post-hyperemia diameter - baseline diameter) / baseline diameter] × 100%. The average of three repeated measurements will be recorded for analysis.
Carotid Corrected Flow Time (CFTc) | Pre-anesthesia measurement.
  Carotid Corrected Flow Time (CFTc) will be measured using Doppler ultrasound at the common carotid artery. The uncorrected carotid flow time will be adjusted for heart rate using Bazett's formula (CFTc = observed flow time / √(R-R interval)). Measurements will be taken preoperatively and at 30 minutes after spinal anesthesia induction. The average of three consecutive measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No